CLINICAL TRIAL: NCT04403412
Title: Short Term Changes of Left Atrial Function and Quality of Life in Patients With Atrial Fibrillation After Left Atrial Appendage Occlusion
Brief Title: Changes of Left Atrial Function and Quality of Life in Patients With Left Atrial Appendage Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruiqin xie (Other)
Responsible Party: Sponsor-Investigator, Ruiqin xie, director of cardiology department, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XierqdoctorLAAO
Record Dates: First submitted 2020-05-03; First posted 2020-05-27 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; left atrial appendage closure; quality of life assessed; left atrial function
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A total of 105 patients with persistent atrial fibrillation(AF), who are persistented more than one year and planned to undergo surgical treatment, will be allocated into two groups. These patients will receive left atrial appendage closure, radiofrequency ablation under the guidance of 3D mapping and left atrial appendage closure combined with radiofrequency ablation, respectively (allocation ratio, 1:1:1).
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers will participate in the operation to record operative parameters such as LA pressure. Other researchers including follow-up personnel and the ultrasonic data analyst are uninformed about the random situation of the patients (patient information is recorded according to the random number. Random numbers corresponding to the random allocation list are stored in the research center. After follow-up of the last patient is completed, the random allocation list is published by the random number designer; and the designer does not participate in the data collection and statistics.)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Left atrial appendage closure group (Experimental)
  Interventions: Procedure: Left atrial appendage closure group
- Radiofrequency ablation group (Experimental)
  Interventions: Procedure: Radiofrequency ablation group
- LAAC combined with radiofrequency ablation group (Experimental)
  Interventions: Procedure: LAAC combined with radiofrequency ablation group

INTERVENTIONS:
Procedure: Left atrial appendage closure group — Left atrial appendage closure Left atrial appendage closure is performed using a single endocardial plug devices guided by fluoroscopic guidance and transesophageal echocardiography
  Arms: Left atrial appendage closure group
Procedure: Radiofrequency ablation group — Radiofrequency ablation Each patient with persistent AF receives circumferential pulmonary vein isolation under the 3D electro-anatomical mapping system , and no additional ablation is performed in the extrapulmonary sites unless the patient is diagnosed with atrial flutter before the operation.
  Arms: Radiofrequency ablation group
Procedure: LAAC combined with radiofrequency ablation group — LAAC combined with radiofrequency ablation group Each patient received the same group of patients with simple radiofrequency ablation radiofrequency ablation treatment at the same time, the transcatheter occlusion of left atrial appendage opening
  Arms: LAAC combined with radiofrequency ablation group

SUMMARY:
A total of 105 patients with atrial fibrillation (AF) are scheduled to receive surgical treatment and will be divided into three groups. Left atrial appendage occlusion (LAAC), three-dimensional mapping guided radiofrequency ablation and LAAC combined radiofrequency ablation (1:1:1) were performed respectively. All patients were examined three-dimensional and two-dimensional ultrasound before operation, 1 and 3 months after operation to measure left atrial (LA) function. The routine blood test and high-sensitivity C-reactive protein were performed in all patients before operation, 1 day and 1 month after operation. B-type natriuretic peptide was detected in all patients before operation and 1 day, 1 month and 3 months after operation. All patients underwent 6-minute walking test and quality of life score before operation, 1 and 3 months after operation.

DETAILED DESCRIPTION:
A total of 105 patients with atrial fibrillation (AF) are scheduled to receive surgical treatment and will be divided into three groups. Left atrial appendage occlusion (LAAC), three-dimensional mapping guided radiofrequency ablation and LAAC combined radiofrequency ablation (1:1:1) were performed respectively. All patients were examined by real-time three-dimensional and two-dimensional ultrasound before operation, 1 and 3 months after operation to measure left atrial (LA) function. All ultrasound data will be stored and the professional director of the ultrasound room will be invited for quantitative analysis. The ultrasound indexes include: left atrial diameter, left atrial ejection fraction, etc. All patients underwent transesophageal echocardiography before operation and 3 months after the operation. Results two experienced ultrasound doctors judged whether there was left atrial thrombus, residual shunt and instrument surface related thrombus. The routine blood test and high-sensitivity C-reactive protein were performed in all patients before operation, 1 day and 1 month after operation. B-type natriuretic peptide was detected in all patients before operation and 1 day, 1 month and 3 months after operation. All patients underwent 6-minute walking test and quality of life score before operation, 1 and 3 months after operation. At the same time, the thickness of crista was measured in all patients. This study will clarify the changes of left atrial function and biochemical quality in patients with AF after LAAC. In addition, this study also observed the effect of radiofrequency ablation combined with LAAC on left atrial function and evaluated whether one-stop surgery has more advantages than simple occlusion or ablation, and analyzed the above results. The patients were followed up for an average of three months to analyze the changes of left atrial function, quality of life and embolism events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AF lasting for more than one year;
2. Antiarrhythmic drugs are ineffective;
3. Age of patients is less than 80 years old;
4. Cha2ds2-vasc score ≥ 2;
5. Not suitable for long-term oral anticoagulants.

Exclusion Criteria:

1. Patients with a history of atrial thrombosis or valvular heart disease (moderate or severe valve stenosis or severe valve regurgitation);
2. Patients undergoing prosthetic heart valve replacement;
3. Pregnant women;
4. Patients with previous liver and kidney diseases, malignant tumors or blood system diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-04-28 (Estimated); Study Completion 2022-04-28 (Estimated)

PRIMARY OUTCOMES:
Left atrial function of postoperative left atrial appendage occlusion detected | 1- 3 month
  Transthoracic ultrasound
changes of 6-minute walking test | 1- 3 month
  6-minute walking test in meter
quality of life assessed | 1- 3 month
  Shot Form 36 Health Survey Questionnaire：the higher the patient's score, the better the quality of life

SECONDARY OUTCOMES:
Residual shunt after transcatheter closure of left atrial appendage detected | 1-3 month
  Transesophageal ultrasound
device-related thrombus after transcatheter closure of left atrial appendage detected | 1-3 month
  Transesophageal ultrasound
C creative protein | 1-3 month
  Blood samples are extracted in all patients to detected
B natriuretic peptide assessed | before and 3 month after operation
  Blood samples are extracted in all patients to detected

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China